CLINICAL TRIAL: NCT07245966
Title: Pharmacokinetics and Pharmacodynamics of High Dose Ceftriaxone in Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sarunyou Chusri, Assoc. Prof. Sarunyou Chusri M.D. Ph.D., Prince of Songkla University
Other Study IDs: REC.66-477-14-1
Record Dates: First submitted 2025-02-21; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As the general treatment method for infectious diseases is to prescribe antibiotics which can be complete at the empirical treatment with the control of the sources of infection, the types of antibiotics that contain the broad spectrum and the proper dose to reduce the severity of infection play an important role. Especially, patients with sepsis should receive antibiotics within 1 hours after the diagnosis since the delay of 1 hour will decrease the rate of survival by 7.6 percent. Ceftriaxone is considered to be Cephalosporin, the antibiotics in the group of β-lactams antibiotic which kills bacteria by preventing the creation of significant cell walls. Ceftriaxone is soluble and can be excreted by the kidney. It is a β-lactams broad spectrum which can kill bacteria broadly including various types of gram-positive and gram-negative. The effectiveness of Ceftriaxone is in accord with the percentage of time that the level of the drug is beyond the minimum inhibitory concentration. According to the research in animals conducted by Craig WA and others, the drug effect to prevent the bacteria growth will occur when the %ft>MIC is more than at least 40%. The rate of prevention will reach the maximal bactericidal effect when the %ft>MIC is equal to 60 to 70%. At the moment, physicians prefer the 60 to 70% of %ft>MIC in the group of Cephalosporins drugs as the main pharmacodynamics to cope with infections.

ELIGIBILITY:
Inclusion Criteria:

* Participants aging over 18 years old with the symptoms of systemic inflammatory response syndrome (SIRS) which requires at least two of the following symptoms
* Temperature over 38 degree Celsius (Fever) or lower than 36 degree Celsius (hypothermia)
* Tachycardia
* Tachypnea, or the detection of PaCO2 under 32 mmHg, or hypocapnia due to hyperventilation
* Participants are about to received Ceftriaxone by the physician
* Weighting equal to or more than 50 kg

Exclusion Criteria:

* Patients with the clinical record of the severe allergy to β-lactam or Ceftriaxone
* Patients received Ceftriaxone within 3 days before the participation
* Having a culture result of being resistant to Ceftriaxone
* Having CLcr lower than 50 ml/min, or receiving hemodialysis, or renal replacement therapy
* Meningitis patients
* Decompensated liver disease
* Pregnant and lactating
* Septic shock patients
* Having the level of serum albumin lower than 2.5 g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 people in total
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Probability of target attainment of the pharmacodynamic index fT>MIC ≥ 100% for ceftriaxone | First 24 hours of ceftriaxone treatment
  The percentage of simulated patients achieving the pharmacodynamic target of free drug time above MIC (fT>MIC ≥ 100%), estimated using population pharmacokinetic modeling incorporating observed plasma concentration-time data and pathogen-specific MIC values or reference MIC distributions.

CONTACTS AND LOCATIONS:
Overall Officials: Sarunyou Chusri, M.D., Ph.D., Principal Investigator — Prince of Songkla University
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No
The data will remain anonymized.